CLINICAL TRIAL: NCT02100982
Title: Developing a Customized Care Intervention to Improve Mental Health Outcomes in Multimorbidity
Brief Title: Improving Communication About Patient Priorities in Multimorbidity
Acronym: ICOM-APP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Marsha Wittink, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MH101236; 5R34MH101236 (NIH)
Record Dates: First submitted 2014-03-19; First posted 2014-04-01 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Chronic Disease
Keywords: Multimorbidity; Communication; Primary Care; Mental Health
MeSH Terms: conditions — Chronic Disease; Communication; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Customized Care (intervention) vs. care as usual
Who Masked: Participant
Masking Description: Participants in both arms use iPad to complete assessments, Customized Care (intervention arm) receives intervention on iPad, care as usual completes assessments only
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Care As Usual (Other): Before the office visit with the PCP, patient participants in the Care As Usual arm will interact with the research staff who will help the participant use an iPad in the waiting room to complete baseline health assessments. Consented patient-participants will be told that the subsequent office visit with the PCP will be audio-recorded to assess patient-PCP communication.
  Interventions: Other: Care As Usual
- Customized Care (Experimental): Before the office visit with the PCP, patient participants in the intervention group will interact with the computer based components of the customized care intervention while in the waiting room. The research staff will help the participant use an iPad in the waiting room and direct them to the Discussion Prioritization tool (DPT). After participants use the DPT, the program automatically generates a customized questions prompt list (QPL) which will be printed out in the office. Study staff will hand the QPL to intervention patients to bring to their office visit with the PCP. Consented patient-participants will be told that the subsequent office visit with the PCP will be audio-recorded to assess patient-PCP communication.
  Interventions: Other: Customized Care

INTERVENTIONS:
Other: Customized Care — Customized Care consists of two components. The first component is a Discussion Prioritization Tool (DPT) which forces patients to make trade-offs between competing concerns to help them determine which are the most important to discuss. The second component is a customized question prompt list (QPL) to help patients communicate their priorities to the PCP. The QPL will be generated after patients use the DPT, and consists of question prompts tailored to the patients' priorities. Consented patient-participants will be told that the subsequent office visit with the PCP will be audio-recorded to assess patient-PCP communication.
  Arms: Customized Care
Other: Care As Usual — Participants in this condition will interact with the research staff who will help the participant use an iPad in the waiting room to complete baseline health assessments. Consented patient-participants will be told that the subsequent office visit with the PCP will be audio-recorded to assess patient-PCP communication.
  Arms: Care As Usual

SUMMARY:
The goal of this study is to develop and test Customized Care, an intervention to help patients dealing with depression and/or anxiety in the context of multiple chronic conditions. Customized Care is designed to help patients communicate about important issues, such as financial and safety concerns, with their primary care providers (PCPs). The intervention will be delivered in patient waiting rooms prior to a routine follow-up visit with the PCP. Phase 1 of the project will ensure that the main components of Customized Care are acceptable to patients and PCPs. Phase 2 will include a pilot study to test the effects of Customized Care on patient-PCP communication.

Participants aged 40 years or older who have a diagnosis of two or more common chronic medical conditions will be recruited from primary care clinics. Patients screening positive for either depression or anxiety will be randomized to Customized Care vs. an active control.

The investigators hypothesize that the Customized Care will improve patient-Primary Care-Provider communication.

DETAILED DESCRIPTION:
Patients with depression or anxiety in the context of multimorbidity (2 or more chronic conditions such as Diabetes, Heart Disease, Arthritis, COPD, Asthma) are often preoccupied with day-to-day concerns related to issues such as finances, safety and functional ability. Determining which issues to discuss, and when to discuss it, is always difficult in the 15-minute primary care visit, but it is especially challenging when patients have multiple diagnoses, symptoms and concerns.

In this application the investigators will develop and test the feasibility of Customized Care, an intervention that capitalizes on decision technology and will be deployed in primary care waiting rooms. The investigators will assess whether customized care will improve outcomes among patients with depression and/or anxiety in the context of multimorbidity. Customized Care consists of two different components designed to improve health outcomes by improving patient-provider communication. The first component is a computer-based discussion prioritization tool (DPT). The DPT forces patients to make trade-offs between competing concerns to help them determine which are the most important to discuss. The second component is a customized question prompt list (QPL) to help patients communicate their priorities to the PCP. The QPL will be generated after patients use the DPT, and consists of question prompts tailored to the patients' priorities.

When patients express their day-to-day concerns, and PCPs become aware of these concerns, the patient-provider alliance can deepen. In addition, patient motivation (perceived autonomy, competence) to manage those everyday concerns and engage in care for chronic disease and associated mental health conditions will increase. This project will lay the ground work for a larger randomized trial to assess whether customized care can improve mental health outcomes among patients with multimorbidity.

The specific aims are:

1. To assess usability of the Customized Care components (the DPT and QPL)
2. To assess feasibility of Customized Care in primary care settings
3. To conduct a pilot study of the effects of Customized Care on patient-PCP communication

ELIGIBILITY:
Inclusion Criteria:

* patients attending a primary care clinic for routine follow-up care
* age 40 or older
* diagnosed with 2 or more chronic medical conditions including: diabetes, heart disease, arthritis, asthma, COPD
* positive screen for symptoms of depression and/or anxiety

Exclusion Criteria:

* non-English speakers
* patients with a diagnosis of dementia or cognitive deficit
* patients with acute medical needs requiring urgent treatment

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-06; Primary Completion 2017-10 (Actual); Study Completion 2018-04-24 (Actual)

PRIMARY OUTCOMES:
Patient-PCP communication | from the beginning to the end of the patient-PCP office visit, average duration of 20 minutes
  After the patient completes the experimental or active comparator intervention on the iPad, the patient will proceed with their office visit. The subsequent conversations between the patient and PCP will be audio-recorded and transcribed. We will use a coding scheme to measure communication during the patient-PCP office visit.

CONTACTS AND LOCATIONS:
Overall Officials: Marsha N Wittink, MD, MBE, Principal Investigator — University of Rochester
Locations (1):
- Highland Family Medicine, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available on request once cleaned and initial analyses by primary team are completed.

REFERENCES:
- [Background] Wittink MN, Yilmaz S, Walsh P, Chapman B, Duberstein P. Customized Care: An intervention to Improve Communication and health outcomes in multimorbidity. Contemp Clin Trials Commun. 2016 Dec 15;4:214-221. doi: 10.1016/j.conctc.2016.10.002. Epub 2016 Oct 11. PMID 28191546
- [Background] Wittink MN, Walsh P, Yilmaz S, Mendoza M, Street RL Jr, Chapman BP, Duberstein P. Patient priorities and the doorknob phenomenon in primary care: Can technology improve disclosure of patient stressors? Patient Educ Couns. 2018 Feb;101(2):214-220. doi: 10.1016/j.pec.2017.08.004. Epub 2017 Aug 8. PMID 28844522